CLINICAL TRIAL: NCT05250011
Title: Early Treatment of Heart Failure: a Non-Interventional Observational Study of Italian Patients With Heart Failure and Initiated on Dapagliflozin
Brief Title: Observation of Italian Patients With Heart Failure Being Treated With Dapagliflozin in Clinical Practice
Acronym: EVOLUTION-HF
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Fullcro s.r.l. (Unknown)
Responsible Party: Sponsor
Other Study IDs: D1699R00030
Record Dates: First submitted 2022-01-20; First posted 2022-02-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure, Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure, Systolic | interventions — dapagliflozin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Single-cohort: Patients initiated on dapagliflozin according to the approved indication for heart failure with reduced ejection fraction (HFrEF) and current medical practice
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin, prescribed as per approved indication and current medical practice. Participants will not receive any experimental disease management intervention or experimental treatment as a consequence of their participation in the study.
  Other Names: Forxiga

SUMMARY:
This is an observational, non-interventional, longitudinal prospective descriptive study including participants diagnosed with Heart Failure with reduced Ejection Fraction (HFrEF) in Italy and initiated on treatment with dapagliflozin according to the approved HFrEF indication. The study is aimed at providing insights into real-world drug utilization and treatment patterns of dapagliflozin in the Italian HFrEF setting, as well as patient-reported outcomes including quality of life.

DETAILED DESCRIPTION:
Heart failure (HF) is a significant burden for public health, affecting more than 63 million people worldwide and expected to increase as the population ages; in Italy, the estimated prevalence of HF is 1-3% and the incidence rate 2-5 cases per 1000 persons per year. Despite advancements in treatment, a HF diagnosis still leads to significant morbidity and mortality and impacts on patients' quality of life (QoL). Dapagliflozin is the first in a novel class of glucose-lowering agents known as sodium-glucose co-transporter-2 (SGLT2) inhibitors, approved for the treatment of Heart Failure with reduced Ejection Fraction (HFrEF). As with all new drugs introduced into clinical practice, there is a strong scientific interest in producing evidence from observational studies regarding the use of dapagliflozin for the treatment of HFrEF in real-world settings with detailed clinical data on heart failure symptoms, outcomes, and health-related QoL.

The overall aim of this observational study is to describe the characteristics of patients in Italy initiating dapagliflozin for the treatment of HFrEF and to provide early insights into real-world dapagliflozin treatment patterns (primary objectives) as well as patient-reported outcomes including quality of life (secondary objectives).

This study is part of a multicountry study programme, including similar studies that will be conducted in other countries with similar objectives. Data from each of the individual studies may be combined in a pooled analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or above 18 years old at the initiation of treatment with dapagliflozin
* Participant received/receiving treatment with dapagliflozin for Heart Failure with reduced Ejection Fraction (HFrEF) in accordance with the approved local dapagliflozin product label, i.e. with an ejection fraction of 40 percent or less
* Signed and dated informed cconsent obtained prior to enrollment into the study

Exclusion Criteria:

* Participant is enrolled less than 14 days or more than 45 days following the initiation of treatment with dapagliflozin
* Prior treatment with dapagliflozin or other treatment with a medicine of the same drug class (sodium-glucose co-transporter-2 - or SGLT2 - inhibitors)
* Initiation of dapagliflozin outside of the approved local dapagliflozin product label for HFrEF
* Diagnosis of Type 1 Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed with dapagliflozin for Heart Failure with reduced Ejection Fraction (HFrEF) according to the approved indication will be eligible for enrollment from both outpatient and inpatient settings.
  The decision to treat a patient with dapagliflozin must be made prior to the decision to enroll the patient. In order to help ensuring this, participants can be enrolled only if they started treatment with dapagliflozin at least 14 days before the enrollment visit, regardless of the treatment being discontinued or suspended in the time between first dapagliflozin prescription and enrollment visit.
  It is expected that 250 participants will be consecutively enrolled in about 11 centres (approximately 23 participants per each study site).
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics of participants | Baseline (enrollment)
  Demographic and clinical characteristics at baseline of study participants
Dapagliflozin treatment pattern | 12 months from prescription of dapagliflozin
  Treatment discontinuation events for dapagliflozin
Other medications treatment patterns | 12 months from prescription of dapagliflozin
  Treatment change events for other medications for heart failure and glucose-lowering medications

SECONDARY OUTCOMES:
Patient Reported Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline (enrollment), Follow-up (3, 6, 12 months after treatment initiation)
  Health-Related Quality of Life: assessment of heart failure symptoms and their impact in terms of physical limitation and quality of life, as captured by the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is scored on a scale from 0 to 100, with higher scores indicating higher quality of life.
Patient Reported Outcome: Medication Adherence Report Scale (MARS-5) | Baseline (enrollment), Follow-up (3, 6, 12 months after treatment initiation)
  Assessment of medication adherence to heart failure treatments, as captured by the five-items version of the Medication Adherence Report Scale (MARS-5). The MARS-5 is scored on a scale from 0 to 25, with higher scores indicating better treatment compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Metra, MD, Principal Investigator — UOC Cardiologia, Spedali Civili di Brescia; Maurizio Volterrani, MD, Principal Investigator — UO Riabilitazione Cardiologica, IRCCS San Raffaele, Roma; Pasquale Perrone Filardi, MD, Principal Investigator — UOC Cardiologia emodinamica e UTIC, Azienda Ospedaliera Universitaria "Federico II", Napoli; Massimo Iacoviello, MD, Principal Investigator — Unità di Cardiologia, Azienda Ospedaliero Universitaria Ospedali Riuniti, Foggia; Pietro Ameri, MD, Principal Investigator — UO Clinica Malattie Apparato Cardiovascolare e UTIC, IRCCS Ospedale Policlinico San Martino, Genova; Andrea Ungar, MD, Principal Investigator — Geriatria UTIG, Azienda Ospedaliero Universitaria Careggi, Firenze; Ciro Indolfi, MD, Principal Investigator — UO Cardiologia-Emodinamica-UTIC, Azienda Ospedaliero Universitaria Mater Domini, Catanzaro; Massimo Volpe, MD, Principal Investigator — UOC Cardiologia, Azienda Ospedaliera Sant'Andrea, Roma; Andrea Mortara, MD, Principal Investigator — Dipartimento di Cardiologia, Policlinico di Monza, Monza; Stefano Carugo, MD, Principal Investigator — Unità di Cardiologia, IRCCS Ca' Granda - Ospedale Maggiore - Policlinico, Milano; Andrea Di Lenarda, MD, Principal Investigator — Cardiologia, Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
Locations (10):
- Italy (10):
  - Research Site, Brescia, BS
  - Research Site, Catanzaro, CZ
  - Research Site, Foggia, FG
  - Research Site, Florence, FI
  - Research Site, Genova, GE
  - Research Site, Monza, MB
  - Research Site, Milan, MI
  - Research Site, Roma, RM
  - Research Site, Trieste, TS
  - Research Site, Napoli

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca sponsored studies via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved, AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1699R00030&attachmentIdentifier=87c18942-4519-441b-8831-b573afd2e3e1&fileName=D1699R00030_Redacted_CSR_Synopsis.pdf&versionIdentifier=